CLINICAL TRIAL: NCT06566508
Title: Effectiveness of Asiaticoside as Intracanal Medication on Infectious/Inflammatory Contents in Teeth With Apical Periodontitis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Salem Abdulrahman Alqahtani, Principal investigator, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A0209023RC
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Intracanal Medication
Keywords: Inflammation; Asiaticoside; Pulpal necrosis
MeSH Terms: conditions — Inflammation; Dental Pulp Necrosis | interventions — Centella asiatica extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calcium Hydroxide (Active Comparator): Intracanal medication
  Interventions: Drug: Calcium Hydroxide Intracanal medication
- Leddermix (Active Comparator): Intracanal medication
  Interventions: Drug: Leddermix Intracanal medication
- Asiaticoside (Active Comparator): Intracanal medication
  Interventions: Drug: Asiaticoside Intracanal medication

INTERVENTIONS:
Drug: Calcium Hydroxide Intracanal medication — Calcium Hydroxide Intracanal medication
  Arms: Calcium Hydroxide
Drug: Leddermix Intracanal medication — Leddermix Intracanal medication
  Arms: Leddermix
Drug: Asiaticoside Intracanal medication — Asiaticoside Intracanal medication
  Other Names: centella asiatica
  Arms: Asiaticoside

SUMMARY:
The objective of this study is to investigate "clinically" the effectiveness of Asiaticoside based intracanal medication compared to the commonly used intracanal medicaments (calcium hydroxide Ca(OH)2 and Ledermix) on the levels of bacteria and inflammatory cytokines in root canals and periradicular tissues of teeth with apical periodontitis.

DETAILED DESCRIPTION:
This study investigate "clinically" the effectiveness of Asiaticoside based intracanal medication compared to the commonly used intracanal medicaments (calcium hydroxide Ca(OH)2 and Ledermix) on the levels of bacteria and inflammatory cytokines in root canals and periradicular tissues of teeth with apical periodontitis.

ELIGIBILITY:
Inclusion Criteria:

• Single-rooted with pulp necrosis and apical periodontitis.

Exclusion Criteria:

Receiving antibiotic treatment within the preceding 3 months.

* Reporting systemic disease.
* Teeth that could not be isolated with rubber dam.
* Teeth with periodontal pockets deeper than 3 mm.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2025-03-03 (Estimated)

PRIMARY OUTCOMES:
counting the number of colonies forming units of bacterial cells Microbiology cell culturing (manual counting technique to the bacterial cells) [Time Frame: up to 7 months] | up to 7 months
  counting the number of colonies forming units of bacterial cells Microbiology cell culturing (manual counting technique to the bacterial cells) [Time Frame: up to 7 months]

SECONDARY OUTCOMES:
using enzyme-linked immunosorbent assay (ELISA test) to measure the amount of Inflammatory Cytokines (TNF-α), (IL-1β) and (PG2) ELISA test to measure the amount of tumor necrotizing factor (TNF-α), interleukin 1β(IL-1β) and prostaglandin E2 (PG2) | up to 25 weeks
  using enzyme-linked immunosorbent assay (ELISA test) to measure the amount of Inflammatory Cytokines (TNF-α), (IL-1β) and (PG2) ELISA test to measure the amount of tumor necrotizing factor (TNF-α), interleukin 1β(IL-1β) and prostaglandin E2 (PG2)

CONTACTS AND LOCATIONS:
Overall Officials: Amany Bader, prof, Study Director — Faculty of Dentistry Mansoura University; Youssry Elhawary, prof, Study Director — Faculty of Dentistry Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Egypt